CLINICAL TRIAL: NCT06234111
Title: Semaglutide and Physical Activity for Obesity and Multimorbidity: Co-designing Healthy Healthcare
Brief Title: Semaglutide and Physical Activity for Obesity and Multimorbidity
Status: Active, not recruiting | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Hoxer Brødsgaard, Principal Investigator, Hvidovre University Hospital
Other Study IDs: F-23061071
Record Dates: First submitted 2024-01-08; First posted 2024-01-31 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Obesity Morbid; Multimorbidity; Obesity
Keywords: Obesity; Multimorbidity; Semaglutide; Glucagon-like peptide-1 receptor agonist; Physical activity; Exercise; Co-design; Patient-centred; Cardiometabolic health; Health-related quality of life; Wegovy
MeSH Terms: conditions — Obesity, Morbid; Obesity; Motor Activity | interventions — semaglutide; Nutrition Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with severe obesity and multimorbidity: Patients with morbid obesity (mainly class II and III) with multiple chronic conditions. Most patients are initially referred for bariatric surgery, but are deemed ineligible for various reasons (typically inability to independently induce weight loss, severe mental disease, eating disorder, and serious comorbidity).
  Interventions: Combination Product: Semaglutide 2.4 mg, total diet replacement, behavioural intervention

INTERVENTIONS:
Combination Product: Semaglutide 2.4 mg, total diet replacement, behavioural intervention — Patients receive a highly specialized interdisciplinary weight loss treatment comprising two phases. Firstly, they engage in a total diet replacement using Nupo for approximately three months to induce a maximal weight loss. After this and for the duration of the entire treatment period, patients receive Semaglutide 2.4 mg and behavioural dietary support to maintain the weight loss and improve health. The total treatment period is two years.
  Other Names: Wegovy; Nupo; Dietary counseling

SUMMARY:
The aim of this observational study is to explore and describe changes in cardiometabolic health, physical activity, physical capacity, and wellbeing during interdisciplinary Semaglutide-based weight loss treatment in patients with severe obesity and multimorbidity.

This study is explorative and therefore does not include hypothesis testing.

DETAILED DESCRIPTION:
This study is part of the project "Semaglutide and Physical Activity for Obesity and Multimorbidity: Co-designing Healthy Healthcare".

While this observational quantitative study aims to provide a comprehensive description of changes in patients' health and wellbeing during and after participation in weight loss treatment, the project also includes a qualitative interview study with a subset of patients from the same population to supplement and expand upon the quantitative findings. Additionally, a smaller subgroup of patients from the same population will eventually be invited to actively contribute to the collaborative development of a physical activity intervention in a co-design process, drawing on insights from the aforementioned studies.

Given its exploratory approach, the study is designed with a flat non-hierarchical outcome structure and multiple evenly valued outcomes measures. This will be reported evenly for all outputs of this research.

ELIGIBILITY:
Study participants are recruited from a particular interdisciplinary weight loss program based at Copenhagen University Hospital Hvidovre. Hence, the study uses the same set of inclusion criteria:

Inclusion criteria:

* Fulfilment of the Danish criteria for bariatric surgery:
* BMI ≥ 35 kg/m2
* Aged ≥ 18 years
* One or more obesity-related conditions (type II diabetes, resistant hypertension, sleep apnea, severe osteoarthritis of the lower extremities)
* One more comorbidities that prevent bariatric surgery

Exclusion criteria are:

* Unwillingness to participate in the study
* Inability to understand Danish
* Cognitive impairments

UPDATE 17.09.2024:

After initiating patient recruitment for the study on 15.02.2024, the project group identified discrepancies between the eligibility criteria and description of the study population as originally reported in the trial registration and those actually applied in the study. As a result, we adjusted both the eligibility criteria and description of the study population in the trial registration on 17.09.2024. These adjustments do not represent a change in the actual patient population but rather offer a more accurate and consistent description of their characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals living in the Capital Region of Denmark can be referred to the weight loss program if they fulfill the Danish criteria for bariatric surgery while having comorbidities that increase the risk of surgery or challenge the accompanying necessary lifestyle changes, thereby making them ineligible for bariatric surgery. Consequently, most patients in the weight loss program are severely burdened by high levels of obesity (usually BMI > 40 kg/m2) and have debilitating somatic and mental multimorbidity (corresponding to Edmonton Obesity Staging System stages 2-4). In other words, patients for whom a substantial and sustained weight loss is expected to lead to tangible and significant health benefits.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Habitual physical activity | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  SENS Motion accelerometry will be used to measure habitual physical activity, defined as time spent non-sedentary and not lying down. We will measure for seven full days. Data will be presented as mean change in hours/day spent physically active between baseline, four months, and follow-up.
  As mentioned, the study is exploratory and designed with a flat outcome hierarchy and multiple evenly valued outcome measures. The registration template requires that one outcome is listed as "primary", which is why this one is listed. This does not mean we consider this outcome more important than other outcomes.

SECONDARY OUTCOMES:
Health-related quality of life: physical | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  The 36-Item Short Form Survey (SF-36) questionaire will be administered for all patients. The physical component summary score and its associated domain scores (physical functioning, role-physical, bodily pain, general health) will be presented as the mean change between baseline, four months, and follow-up scores. Possible scores range from 0 to 100, with higher scores indicating better health status.
10-years cardiovascular risk (previous cardiovascular disease) | Baseline (± 2 weeks), 4 months (± 2 weeks) and 21 months (± 2 weeks).
  The 10-years risk of myocardial infarction, stroke or cardiovascular death wil be calculated using the SMART risk assessment tool. This specific risk assessment tool will be used only for individuals with previous cardiovascular disease, as it was designed for this particular population. All data needed for the SMART risk assessment tool are already being collected as routine practice. Results derived from the three different risk assessment tools will be combined, as they measure the exact same outcome (10-years cardiovascular risk). They will be presented as mean change in absolute risk between baseline, four months, and follow-up.
10-years cardiovascular risk (type 2 diabetes) | Baseline (± 2 weeks), 4 months (± 2 weeks) and 21 months (± 2 weeks).
  The 10-years risk of myocardial infarction, stroke or cardiovascular death wil be calculated using the ADVANCE risk assessment tool. This specific risk assessment tool will be used for individuals with type 2 diabetes and without previous cardiovascular disease, as it was designed for this particular population. All data needed for the ADVANCE risk assessment tool are already being collected as routine practice. Results derived from the three different risk assessment tools will be combined, as they measure the exact same outcome (10-years cardiovascular risk). They will be presented as mean change in absolute risk between baseline, four months, and follow-up.
10-years cardiovascular risk (apparently healthy) | Baseline (± 2 weeks), 4 months (± 2 weeks) and 21 months (± 2 weeks).
  The 10-years risk of myocardial infarction, stroke or cardiovascular death wil be calculated using the SCORE2 risk assessment tool. This specific risk assessment tool will be used for individuals without type 2 diabetes and previous cardiovascular disease, as it was designed for this particular population. All data needed for the SCORE2 risk assessment tool are already being collected as routine practice. Results derived from the three different risk assessment tools will be combined, as they measure the exact same outcome (10-years cardiovascular risk). They will be presented as mean change in absolute risk between baseline, four months, and follow-up.

OTHER OUTCOMES:
Body weight | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  The patients' body weight will be measured and presented as mean percentual change in weight between baseline, four months, and follow-up.
Waist circumference | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  Waist circumference will be measured in cm with 1 decimal with a tape measurer and presented as mean change between baseline, four months, and follow-up.
Health-related quality of life: mental | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  The 36-Item Short Form Survey (SF-36) questionaire will be administered for all patients. The mental component summary score and its associated domain scores (vitality, social functioning, role-emotional, mental health) will be presented as the mean change between baseline, four months, and follow-up scores. Possible scores range from 0 to 100, with higher scores indicating better health status.
Weight bias internalization | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  The Weight Bias Internalization Scale (WBIS) will be administered for all patients. The WBIS includes 19-items to be rated on a 7-point Likert scale ranging from "strongly disagree" to "strongly agree". The mean score of all 19 items will be calculated and presented as mean change between baseline, four months, and follow-up. Possible mean scores range from 1 to 7, with higher scores indicating greater weight bias internalization.
Cardiorespiratory fitness | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  Maximal oxygen uptake (VO2max) will be measured with the "Seismofit System". The Seismofit sensor is placed on the sternum, where it measures seismocardiography (the vibrations generated by the heart and transmitted through the chest). These measures are coupled with information on sex, age, weight, and height. Using an algorithm, the Seismofit System then estimates VO2max. Change in VO2max will be presented as mean change between baseline, four months, and follow-up.
Lower body strength | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  Lower body strength and endurance will be measured with the 30-Seconds Sit-To-Stand test and will be presented as mean change in repetitions between baseline, four months, and follow-up.
Walking capacity and endurance | Baseline (± 2 weeks), 4 months (± 2 weeks) and 24 months (± 2 weeks).
  Walking capacity and endurance will be measured with the 6-Minute Walk Test and will be presented as mean change in meters walked between baseline, four months, and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus H Brødsgaard, MSc, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No